CLINICAL TRIAL: NCT05203185
Title: Nudging Provider Adoption of Clinical Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-01316; 5K23HL145114-02 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Embolism
Keywords: Clinical Decision Support; Pulmonary Embolism; Behavioral Design; Health Informatics
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Site (Experimental): Full time employed Emergency Department providers will use the new CDS tool, Pulmonary Embolism Risk Kalculator (PERK), which includes nudges to improve use and will be integrated into the electronic medical record and will be accessible for 6 months
  Interventions: Other: Pulmonary Embolism Risk Kalculator (PERK)
- No Intervention Site (No Intervention): Full time employed Emergency Department providers used a CDS tool, Pulmonary Embolism Calculator (PE CALC), without nudges to improve use, to reduce unnecessary imaging in the diagnosis of pulmonary embolism (PE) in the emergency department (ED).

INTERVENTIONS:
Other: Pulmonary Embolism Risk Kalculator (PERK) — Nudges are applications of behavioral science, defined as positive reinforcement and indirect suggestions that have a non-forced effect on decision making. Nudges will be to the PE CALC CDS tool to develop the new CDS tool, PERK.
  Arms: Intervention Site

SUMMARY:
The central hypothesis of this proposal is that the addition of a theory-informed "nudge" to a clinical decision support (CDS) tool will address identified behavioral barriers to use and significantly improve adoption by providers. Nudges are applications of behavioral science, defined as positive reinforcement and indirect suggestions that have a non-forced effect on decision making. This study will use a behavioral theory-informed process to develop a new CDS tool that includes a nudge that addresses barriers to adoption.

DETAILED DESCRIPTION:
The research team developed and pilot tested two CDS tools for pulmonary embolism (PE) risk stratification in the Emergency Department (ED). One of the tools incorporated two behavioral theory-informed nudges in the user interface. The research team's objective was to pilot test the tools to demonstrate feasibility as well as examine preliminary efficacy of the nudges on provider adoption of the tool. This cluster non-randomized controlled trial took place between September 20th, 2021 and March 3rd, 2022 in two EDs that are a part of a large academic health system in the New York City metropolitan area. All ED providers (physicians, physician assistants and nurse practitioners) seeing patients for the evaluation of PE during this time were included in the trial. The EDs were chosen based on their comparable size and acuity levels.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors, nurse practitioners and physician assistants working full time at Huntington Hospital and Long Island Jewish Valley Stream

Exclusion Criteria:

* Does not meet the inclusion criteria

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1612 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Safiya Richardson, MD, MPH, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Huntington Hospital, Huntington, New York
  - Long Island Jewish Valley Stream, Valley Stream, New York

REFERENCES:
- [Derived] Richardson S, Dauber-Decker KL, Solomon J, Seelamneni P, Khan S, Barnaby DP, Chelico J, Qiu M, Liu Y, Sanghani S, Izard SM, Chiuzan C, Mann D, Pekmezaris R, McGinn T, Diefenbach MA. Effect of a behavioral nudge on adoption of an electronic health record-agnostic pulmonary embolism risk prediction tool: a pilot cluster nonrandomized controlled trial. JAMIA Open. 2024 Aug 1;7(3):ooae064. doi: 10.1093/jamiaopen/ooae064. eCollection 2024 Oct. PMID 39091509

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Site - Providers: Providers at the site assigned to the intervention:
  Full time employed Emergency Department providers will use the new CDS tool, Pulmonary Embolism Risk Kalculator (PERK), which includes nudges to improve use and will be integrated into the electronic medical record and will be accessible for 6 months
  Pulmonary Embolism Risk Kalculator (PERK): Nudges are applications of behavioral science, defined as positive reinforcement and indirect suggestions that have a non-forced effect on decision making. Nudges will be to the PE CALC CDS tool to develop the new CDS tool, PERK.
- No Intervention Site - Providers: Providers at the site assigned to no intervention:
  Full time employed Emergency Department providers used a CDS tool, Pulmonary Embolism Calculator (PE CALC), without nudges to improve use, to reduce unnecessary imaging in the diagnosis of pulmonary embolism (PE) in the emergency department (ED).
- Intervention Site - Patients: Patients at the site assigned to the intervention:
  Full time employed Emergency Department providers will use the new CDS tool, Pulmonary Embolism Risk Kalculator (PERK), which includes nudges to improve use and will be integrated into the electronic medical record and will be accessible for 6 months
  Pulmonary Embolism Risk Kalculator (PERK): Nudges are applications of behavioral science, defined as positive reinforcement and indirect suggestions that have a non-forced effect on decision making. Nudges will be to the PE CALC CDS tool to develop the new CDS tool, PERK.
- No Intervention Site - Patients: Patients at the site assigned to no intervention:
  Full time employed Emergency Department providers used a CDS tool, Pulmonary Embolism Calculator (PE CALC), without nudges to improve use, to reduce unnecessary imaging in the diagnosis of pulmonary embolism (PE) in the emergency department (ED).
Period: Overall Study
Arm/Group | Intervention Site - Providers | No Intervention Site - Providers | Intervention Site - Patients | No Intervention Site - Patients
Started | 49 | 35 | 793 | 735
Completed | 49 | 35 | 793 | 735
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sex, ethnicity and race data were not collected from Provider participants. Sex data were not collected from Patient participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Site - Providers | No Intervention Site - Providers | Intervention Site - Patients | No Intervention Site - Patients | Total
Number analyzed (Participants) | 49 | 35 | 793 | 735 | 1612
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [33 to 44] | 35 [33 to 38] | 65 [53 to 79] | 64 [49 to 77] | 51 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data were not collected from study participants.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data were not collected from Provider participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 793 | 735 | 1528
    Hispanic or Latino |  |  | 69 | 32 | 101
    Not Hispanic or Latino |  |  | 673 | 617 | 1290
    Unknown or Not Reported |  |  | 51 | 86 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data were not collected from Provider participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 793 | 735 | 1528
    American Indian or Alaska Native |  |  | 0 | 0 | 0
    Asian |  |  | 14 | 32 | 46
    Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Black or African American |  |  | 42 | 435 | 477
    White |  |  | 618 | 146 | 764
    More than one race |  |  | 0 | 0 | 0
    Unknown or Not Reported |  |  | 119 | 122 | 241
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 35 | 793 | 735 | 1612

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patient Visits Where the Provider Adopted the Pulmonary Embolism Risk Kalculator (PERK) Tool
Description: The tool is considered adopted during a patient visit if the provider accepted the recommendation given by the PERK tool (i.e., a D-dimer was recommended and ordered or a CT pulmonary angiogram (CTPA) was recommended and ordered). This outcome measure is assessed using electronic health record (EHR) data from the patient visit.
Time Frame: Up to Month 6
Measure: Number; unit: Percentage of Patient Visits
Units Other Than Participants: Patient Visits
Groups:
- Intervention Site - Patients and Providers: Patients and Providers at the site assigned to the intervention:
  Full time employed Emergency Department providers will use the new CDS tool, Pulmonary Embolism Risk Kalculator (PERK), which includes nudges to improve use and will be integrated into the electronic medical record and will be accessible for 6 months
  Pulmonary Embolism Risk Kalculator (PERK): Nudges are applications of behavioral science, defined as positive reinforcement and indirect suggestions that have a non-forced effect on decision making. Nudges will be to the PE CALC CDS tool to develop the new CDS tool, PERK.
- No Intervention Site - Patients and Providers: Patients and Providers at the site assigned to no intervention:
  Full time employed Emergency Department providers used a CDS tool, Pulmonary Embolism Calculator (PE CALC), without nudges to improve use, to reduce unnecessary imaging in the diagnosis of pulmonary embolism (PE) in the emergency department (ED).
Arm/Group | Intervention Site - Patients and Providers | No Intervention Site - Patients and Providers
Number analyzed (Participants) | 842 | 770
Number analyzed (Patient Visits) | 793 | 735
Percentage of Patient Visits | 39.11 | 20.66

2. Secondary Outcome: Percentage of PE-Designated CTPA Tests That Are Positive for PE
Description: Monitored using EHR reporting data. Calculated as the percentage of CTPA tests ordered to evaluate for PE that are positive for PE.
Time Frame: Up to Month 6
Measure: Number; unit: Percentage of PE-Designated CTPA Tests
Units Other Than Participants: PE-Designated CTPA Tests
Arm/Group | Intervention Site - Patients and Providers | No Intervention Site - Patients and Providers
Number analyzed (Participants) | 842 | 770
Number analyzed (PE-Designated CTPA Tests) | 707 | 641
Percentage of PE-Designated CTPA Tests | 26.45 | 10.76

ADVERSE EVENTS:
Time Frame: 6 months.
Description: PI reviewed EHR reporting data every two weeks during the study. Adverse events, serious adverse events, and all-cause mortality data were not collected from Provider participants; Provider participant arms are not included below.
Arm/Group | Intervention Site - Patients | No Intervention Site - Patients
All-Cause Mortality (participants affected / at risk) | 0/793 | 0/735
Serious Adverse Events (participants affected / at risk) | 0/793 | 0/735
Other Adverse Events (participants affected / at risk) | 0/793 | 0/735

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT05203185/Prot_SAP_000.pdf